CLINICAL TRIAL: NCT06301334
Title: Block and Erector Comparative Study Between Costotransverse Spinae Plane Block for Postoperative Analgesia in Patients Undergoing Thoracotomy
Brief Title: Block and Erector Comparative Study Between Costotransverse Spinae Plane Block in Patients Undergoing Thoracotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mokhtar Ahmed, Resident of anesthesia department, Sohag university hospital, Sohag University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-01-11MS
Record Dates: First submitted 2024-02-14; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Pain Mangement of Thoracotomy
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group CTB (Active Comparator): n=30): patients included in this group will receive unilateral US-guided CTB after general anesthesia. The CTB will be performed by using 20 ml bupivacaine 0.25%
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution
- Group ESPB (Active Comparator): patients included in this group will receive unilateral US-guided ESPB after general anesthesia. The ESB will be performed by using 20 ml bupivacaine 0.25%
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution

INTERVENTIONS:
Drug: Bupivacaine 0.25% Injectable Solution — Group CTB (n=30): patients included in this group will receive unilateral US-guided CTB after general anesthesia. The CTB will be performed by using 20 ml bupivacaine 0.25% Group ESPB (n=30): patients included in this group will receive unilateral US-guided ESPB after general anesthesia. The ESB will be performed by using 20 ml bupivacaine 0.25%

SUMMARY:
A thoracotomy requires a very painful incision, involving multiple muscle layers, rib resection and continuous motion as the patient breathes. Treatment of acute post thoracotomy pain is particularly important not only to keep the patient comfortable but also to minimize pulmonary complications

Though epidural analgesia was once considered as the gold standard for post-thoracotomy pain management, it is not recommended for pain control after thoracotomy surgery because it is associated with high potential risks of dural puncture, nerve lesions, epidural hematoma and hypotension(4). Thoracic paravertebral block (TPVB) and intercostal nerve block are well described and recognized techniques for postoperative analgesia following thoracic surgeries, such as thoracotomy and mastectomy

ELIGIBILITY:
Inclusion Criteria:

* • Age from 18 to 75 years old.

  * Both sexes.
  * American Society of Anesthesiologists (ASA) physical status I-II-III.
  * Patient undergoing unilateral thoracotomy surgery.

Exclusion Criteria:

* • BMI more than 30 kg/m2.

  * Patients who are taking analgesics for chronic illness or have a history of substance abuse.
  * Patients who are unable to describe their postoperative pain (e.g., language barrier or neuropsychiatric disorder).
  * Patients with a history of coagulopathy.
  * Severe heart diseases.
  * Hepatic or renal insufficiency.
  * Infection at the site of infiltration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
study aims to compare the analgesic efficacy of CTB and ESPB for post-operative analgesia in patients undergoing thoracotomy. | 5months
  study aims to compare the analgesic efficacy of CTB and ESPB for post-operative analgesia in patients undergoing thoracotomyA standardized analgesic regimen will be prescribed in the post-operative period. All patients will receive paracetamol 1 gm every 6 h as routine analgesia. If visual analogue scale (VAS) is more than 3, intravenous morphine 3mg will be administered as rescue analgesia If visual analogue scale (VAS) is more than 5

SECONDARY OUTCOMES:
The secondary outcome is the total postoperative morphine consumption, time of first analgesic, | 5months
  The secondary outcome is the total postoperative morphine consumption, time of first analgesic A standardized analgesic regimen will be prescribed in the post-operative period. All patients will receive paracetamol 1 gm every 6 h as routine analgesia. If visual analogue scale (VAS) is more than 3, intravenous morphine 3mg will be administered as rescue analgesia If visual analogue scale (VAS) is more than 5

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mijatovic D, Bhalla T, Farid I. Post-thoracotomy analgesia. Saudi J Anaesth. 2021 Jul-Sep;15(3):341-347. doi: 10.4103/sja.SJA_743_20. Epub 2021 Jun 19. PMID 34764841
- [Background] Liu Y, Xiao S, Yang H, Lv X, Hou A, Ma Y, Jiang Y, Duan C, Mi W; CAPOPS Group. Postoperative pain-related outcomes and perioperative pain management in China: a population-based study. Lancet Reg Health West Pac. 2023 Jun 10;39:100822. doi: 10.1016/j.lanwpc.2023.100822. eCollection 2023 Oct. PMID 37927993
- [Background] Singariya G, Kamal M, Paliwal B. Pain after thoracotomy: Conquered or to be conquered? Indian J Anaesth. 2023 Feb;67(Suppl 1):S12-S14. doi: 10.4103/ija.ija_90_23. Epub 2023 Feb 10. No abstract available. PMID 37065951
- [Background] Huang W, Wang W, Xie W, Chen Z, Liu Y. Erector spinae plane block for postoperative analgesia in breast and thoracic surgery: A systematic review and meta-analysis. J Clin Anesth. 2020 Nov;66:109900. doi: 10.1016/j.jclinane.2020.109900. Epub 2020 Jun 2. PMID 32502778